CLINICAL TRIAL: NCT06781827
Title: Application Research of Lactobacillus Reuteri in the Treatment of Inflammatory Bowel
Brief Title: Research on the Use of Probiotics in the Prevention and Treatment of Inflammatory Bowel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WK20250106
Record Dates: First submitted 2025-01-10; First posted 2025-01-17 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Daily intervention with Limosilactobacillus reuteri LR08 (10 billion CFU, 2g) for 8 weeks, stored in a cool and dry place.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Every day to give 3 g maltodextrin intervention for 8 weeks. Store in a cool and dry place.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of the study lasts 8 weeks and each patient will be visited 4 times (January, March, June, and December).
  Arms: Probiotic
Dietary Supplement: Maltodextrin — The experimental phase of this study had last 8 weeks and each patient will make 4 visits (January, March, June, and December).
  Arms: Placebo

SUMMARY:
This project involves the use of oral Lactobacillus reuteri as an adjunct therapy for 8 weeks. Endoscopic observation of intestinal inflammation will be conducted at 1 month, 3 months, 6 months, and 12 months after the administration of the drug. Intestinal fluid will be collected endoscopically for 16S RNA analysis to assess changes in the gut microbiota. Inflammatory changes in the patients will be detected through peripheral blood tests, and fecal calprotectin levels will be measured to evaluate the progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Be over 18 years old
2. Agree to sign informed consent; Have been diagnosed with IBD for at least 3 months but not more than 3 years -

Exclusion Criteria:

1. Does not meet the diagnostic criteria of CD
2. Patients with other autoimmune diseases, infectious diseases and malignant tumors Patients with CD during pregnancy and lactation; Patients with serious diseases of the liver, kidney, heart and lung, etc
3. Patients with allergic diseases such as asthma and allergic rhinitis; alcoholic Patients with mental illness
4. Patients with suspected cancer in their intestines
5. Antibiotics, probiotics and prebiotics have been used in the past three months Had intestinal surgery (except appendicitis surgery)
6. There is currently an infection
7. He has had cancer in the last 5 years -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of Intestinal Inflammation Assessed by Endoscopic Scoring System | 12 months
  The intestinal inflammation will be assessed using the Endoscopic Scoring System, which will be observed under endoscope at 1 month, 3 months, 6 months, and 12 months after the administration of the drug.

SECONDARY OUTCOMES:
Assessment of Intestinal Flora Changes Using 16S RNA Analysis | 8 weeks
  Part of the intestinal fluid was collected under endoscope, and 16S RNA analysis was conducted to evaluate the changes in the intestinal flora composition.
Assessment of Inflammatory Changes Using Peripheral Blood Inflammatory Markers | 8 weeks
  The inflammatory changes were detected by analyzing peripheral blood for specific inflammatory markers such as C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), and other relevant cytokines.
Disease progression | 8 weeks
  The progress of the disease was assessed by collecting fecal samples to detect the change of calcarein
Evaluation of Crohn's Disease Severity Using the Crohn's Disease Activity Index (CDAI) | 8 weeks
  The Crohn's Disease Activity Index (CDAI) was used to evaluate the disease severity of CD. The CDAI score ranges from 0 to 600, with higher scores indicating more severe disease. The index is calculated by combining the daily frequency of bowel movements, abdominal pain score (0-10), general well-being (0-7), and the presence of abdominal mass (0-2). Additionally, the Simple Endoscopic Score for Crohn's Disease (SES-CD) was used for endoscopic scores, which ranges from 0 to 42, with higher scores indicating more severe endoscopic findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Department of Jiangsu Province （Suqian）Hospital, Suqian, Jiangsu, China